CLINICAL TRIAL: NCT01006837
Title: Hypothermia in the Trauma Patient - Temperature Changes During Transport and Initial Treatment in Hospital
Brief Title: Hypothermia in the Trauma Patient - When do Trauma Patients Get Cold?
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/1263 (REK)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Hypothermia
Keywords: trauma patients; severe injury; ISS ≥9
MeSH Terms: conditions — Hypothermia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze changes in core body- and skin temperature during pre-hospital and early in-hospital treatment of multi-traumatized patients. The researchers want to investigate when trauma patients get cold and to what extent.

DETAILED DESCRIPTION:
Hypothermia is a common finding in severely traumatized patients. Decreases in core temperature during the course of initial evaluation and resuscitation are common, and can contribute to poor outcomes in multi-traumatized patients.

In this study the temperature will be recorded continually with multiple skin probes and an ear-probe from the site of the accident to arrival in the intensive care unit (including time in primary surgery, if any).

ELIGIBILITY:
Inclusion Criteria:

* trauma patient with a ISS 9 or above.

Exclusion Criteria:

* <12 years old

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients transported to St. Olavs Hospital (Trondheim, Norway), followed by an anesthesiologist from the norwegian air ambulance and taken care of by the trauma team in the emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Survival to discharge | one year

SECONDARY OUTCOMES:
Degree of hypothermia | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Skogvoll, MD, PhD, Study Chair — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, department of anesthesia, Trondheim, Norway

REFERENCES:
- [Result] Uleberg O, Eidstuen SC, Vangberg G, Skogvoll E. Temperature measurements in trauma patients: is the ear the key to the core? Scand J Trauma Resusc Emerg Med. 2015 Nov 19;23:101. doi: 10.1186/s13049-015-0178-z. PMID 26585382